CLINICAL TRIAL: NCT01521871
Title: A Prospective, Randomised Study on Tissue Glue (Cyanoacrylate) Versus Conventional Suture for Skin Closure in Laparoscopic Living Donor Nephrectomy
Brief Title: Tissue Glue (Cyanoacrylate) Versus Conventional Suture in Kidney Donors
Acronym: TG-CYANO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Ole Morten Øyen, Principal Investigator, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 214603
Record Dates: First submitted 2012-01-12; First posted 2012-01-31 (Estimated); Results first posted 2014-11-04 (Estimated); Last update posted 2014-11-04 (Estimated); Status verified 2014-11

CONDITIONS: Skin Closure of Surgical Incisions by Tissue Glue vs Suture
Keywords: Tissue glue; Cyanoacrylate; Wound closure; Living donor nephrectomy; Surgical wound closure
MeSH Terms: interventions — Bandages

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tissue glue wound closure (Experimental): Skin wound closure by tissue glue
  Interventions: Procedure: Skin wound closure by tissue glue
- Conventional suture + dressing (Active Comparator): Skin wound closure by conventional suture + dressing
  Interventions: Procedure: Skin wound closure by conventional suture + dressing

INTERVENTIONS:
Procedure: Skin wound closure by tissue glue — The glue is used both as closure device and as wound dressing.
  Other Names: CE-marked Liquiband Laparoscopic/Surgical: CE 0123
  Arms: Tissue glue wound closure
Procedure: Skin wound closure by conventional suture + dressing — Suture: Intracutaneous skin closure, by running, absorbable suture (Caprosyn 4-0) Dressing: Conventional textile dressing (Mepor)
  Arms: Conventional suture + dressing

SUMMARY:
By means of a prospective, randomised trial the investigators want to examine skin closure in living donors - subjected to laparoscopic, hand-assisted nephrectomy - by tissue glue (Cyanoacrylate (Liquiband)) versus conventional, intracutaneous suture and dressing (1 : 1; 30 + 30 donors).

Study hypothesis: (i) Latest generation tissue glue (Cyanoacrylate (Liquiband)) is at least as good as conventional suture regarding wound healing/complications. (ii) Peroperatively, tissue glue is faster than conventional suture.

DETAILED DESCRIPTION:
At Oslo University Hospital Rikshospitalet, the principal investigator have since 1998 been involved in developing minimally invasive techniques for living donor nephrectomy (LDN). Since 2009 all LDN's have been performed by laparoscopic, hand-assisted technique; by means of 'handport' and 3 laparoscopic ports (5/12 mm).

The investigators consider use of tissue glue instead of suture as another small step towards less invasive surgery.

Since 2000 there has been many reports, and even Cochrane reviews on the use/safety of tissue glue for skin closure. However, very few randomised studies have been performed with the latest generation tissue glue; Cyanoacrylate, with a critical mixture of octyl-:butyl-acrylate. And in Norway there has been no research in this field.

On this basis, the investigators intend to examine skin closure in living donors, a very healthy/homogenous study population, subjected to laparoscopic, hand-assisted nephrectomy, by a prospective, randomised trial: Tissue glue (Cyanoacrylate (Liquiband)) versus conventional, intracutaneous suture and dressing (1 : 1; 30 + 30 donors).

Primarily, the investigators will examine wound healing/complications by wound observation at postop. days 2 + 4 + 'at departure', with numerical scales for secretion, gaps, edema, rubor - as well as infection/bacteriology and complications/ reinterventions. In addition, the donors' self-satisfaction with the wound handling will be registered. Furthermore, the investigators will look at time consumption during surgery, price, stay in hospital and cosmesis judged at 2-3 months postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Living kidney donor with informed consent
* Approved comprehensive work-up/evaluation at local hospital

Exclusion Criteria:

* Allergy towards acrylate or similar chemicals
* Unable to communicate in norwegian language

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2012-01; Primary Completion 2012-11 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ole M Øyen, MD, PhD, Principal Investigator — Oslo University Hospital; Morten Skauby, MD, Study Chair — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Rikshospitalet, Clinic for Cancer, Surgery and Transplantation, Dep. for Transplantation Medicine, Oslo, Oslo County, Norway

REFERENCES:
- [Background] Blondeel PN, Murphy JW, Debrosse D, Nix JC 3rd, Puls LE, Theodore N, Coulthard P. Closure of long surgical incisions with a new formulation of 2-octylcyanoacrylate tissue adhesive versus commercially available methods. Am J Surg. 2004 Sep;188(3):307-13. doi: 10.1016/j.amjsurg.2004.04.006. PMID 15450839
- [Background] Dowson CC, Gilliam AD, Speake WJ, Lobo DN, Beckingham IJ. A prospective, randomized controlled trial comparing n-butyl cyanoacrylate tissue adhesive (LiquiBand) with sutures for skin closure after laparoscopic general surgical procedures. Surg Laparosc Endosc Percutan Tech. 2006 Jun;16(3):146-50. doi: 10.1097/00129689-200606000-00005. PMID 16804456
- [Background] Farion K, Osmond MH, Hartling L, Russell K, Klassen T, Crumley E, Wiebe N. Tissue adhesives for traumatic lacerations in children and adults. Cochrane Database Syst Rev. 2002;2002(3):CD003326. doi: 10.1002/14651858.CD003326. PMID 12137689
- [Background] Coulthard P, Esposito M, Worthington HV, van der Elst M, van Waes OJ, Darcey J. Tissue adhesives for closure of surgical incisions. Cochrane Database Syst Rev. 2010 May 12;(5):CD004287. doi: 10.1002/14651858.CD004287.pub3. PMID 20464728
- [Background] Liversedge NH. Get Stuck In! Hands On Experiences With Surgical Skin Glue. Obs & Gynae Product News 2007; Issue 14: 24-28

RESULTS

PARTICIPANT FLOW:
Groups:
- Conventional Suture + Dressing: Skin wound closure by conventional suture + dressing
  Skin wound closure by conventional suture + dressing : Suture: Intracutaneous skin closure, by running, absorbable suture (Caprosyn 4-0) Dressing: Conventional textile dressing (Mepor)
- Tissue Glue Wound Closure: Skin wound closure by tissue glue
  Skin wound closure by tissue glue : The glue is used both as closure device and as wound dressing.
Period: Overall Study
Arm/Group | Conventional Suture + Dressing | Tissue Glue Wound Closure
Started | 32 | 32
Completed | 32 | 32
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Conventional Suture + Dressing | Tissue Glue Wound Closure | Total
Number analyzed (Participants) | 32 | 32 | 64
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 32 | 26 | 58
  >=65 years | 0 | 6 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.4 (11.25) | 48.4 (13.58) | 47.9 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 22 | 38
  Male | 16 | 10 | 26
Region of Enrollment [Number; unit: participants]
  Norway | 32 | 32 | 64

OUTCOME MEASURES:

1. Primary Outcome: Wound Healing by Numerical Scales for Rubor Postoperative Day 2.
Description: The evaluation is performed by the use of a previously set numerical scale for rubor (0-3; 0: pale, 3: typically infectious). Both arms/groups are evaluated day 2 postoperatively to measure any difference between the two skin closure methods. A high score is used as indicator of traumaticity towards the skin and a higher potential for wound infection.
Time Frame: At postoperative day 2 (2 days after kidney donation)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tissue Glue Wound Closure | Conventional Suture + Dressing
Number analyzed (Participants) | 32 | 32
units on a scale | 0.516 (0.311) | 0.984 (0.364)

2. Primary Outcome: Wound Healing by Numerical Scales for Rubor Postoperative Day 4.
Description: The evaluation is performed by the use of a previously set numerical scale for rubor (0-3; 0: pale, 3: typically infectious). Both arms/groups are evaluated day 4 postoperatively to measure any difference between the two skin closure methods. A high score is used as indicator of traumaticity towards the skin and a higher potential for wound infection.
Time Frame: At postop. day 4 (4 days after kidney donation)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tissue Glue Wound Closure | Conventional Suture + Dressing
Number analyzed (Participants) | 32 | 32
units on a scale | 0.547 (0.261) | 0.750 (0.335)

3. Primary Outcome: Wound Healing by Numerical Scales for Rubor at Discharge From Hospital.
Description: as for outcome 2
Time Frame: At departure from Surgical Dep. to the patients home, usually at postop. day 4, 5, 6 or 7
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tissue Glue Wound Closure | Conventional Suture + Dressing
Number analyzed (Participants) | 32 | 32
units on a scale | 0.476 (0.288) | 0.639 (0.279)

4. Primary Outcome: Wound Healing by Numerical Scales for Secretion Postoperative Day 2.
Description: The evaluation is performed by the use of a previously set numerical scale for secretion ((0-3; 0: totally dry - 3: continuous secretion). Both arms/groups are evaluated day 2 postoperatively to measure any difference between the two skin closure methods. A high score is used as indicator of traumaticity towards the skin and a higher potential for wound infection.
Time Frame: Postop. day 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tissue Glue Wound Closure | Conventional Suture + Dressing
Number analyzed (Participants) | 32 | 32
units on a scale | 0.328 (0.478) | 0.594 (0.384)

5. Primary Outcome: Wound Healing by Numerical Scales for Secretion Postoperative Day 4.
Description: The evaluation is performed by the use of a previously set numerical scale for secretion ((0-3; 0: totally dry - 3: continuous secretion). Both arms/groups are evaluated day 4 postoperatively to measure any difference between the two skin closure methods. A high score is used as indicator of traumaticity towards the skin and a higher potential for wound infection.
Time Frame: Postop. day 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tissue Glue Wound Closure | Conventional Suture + Dressing
Number analyzed (Participants) | 32 | 32
units on a scale | 0.375 (0.484) | 0.117 (0.275)

6. Primary Outcome: Wound Healing by Numerical Scales for Secretion at Discharge From Hospital.
Description: as for outcome 5
Time Frame: At departure from Surgical Dep. to the patients home, usually at postop. day 4, 5, 6 or 7
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tissue Glue Wound Closure | Conventional Suture + Dressing
Number analyzed (Participants) | 32 | 32
units on a scale | 0.286 (0.396) | 0.028 (0.115)

7. Primary Outcome: Wound Healing by Numerical Scales for Oedema Postoperative Day 2.
Description: The evaluation is performed by the use of a previously set numerical scale for oedema (0-1; 0: no elevation - 1: oedema causing > 2 mm elevation). Both arms/groups are evaluated day 2 postoperatively to measure any difference between the two skin closure methods. A high score is used as indicator of traumaticity towards the skin and a higher potential for wound infection.
Time Frame: Postop. day 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tissue Glue Wound Closure | Conventional Suture + Dressing
Number analyzed (Participants) | 32 | 32
units on a scale | 0 (0) | 0.094 (0.292)

8. Primary Outcome: Wound Healing by Numerical Scales for Oedema Postoperative Day 4.
Description: as for outcome 7
Time Frame: Postop. day 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tissue Glue Wound Closure | Conventional Suture + Dressing
Number analyzed (Participants) | 32 | 32
units on a scale | 0 (0) | 0.083 (0.227)

9. Primary Outcome: Wound Healing by Numerical Scales for Oedema at Discharge From Hospital.
Description: as for outcome 7
Time Frame: At departure from Surgical Dep. to the patients home, usually at postop. day 4, 5, 6 or 7
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tissue Glue Wound Closure | Conventional Suture + Dressing
Number analyzed (Participants) | 32 | 32
units on a scale | 0 (0) | 0.111 (0.266)

10. Primary Outcome: Wound Healing by Numerical Scales for Blisters Postoperative Day 2.
Description: The evaluation is performed by the use of a previously set numerical scale for blisters (0: none - 3: abundant). Both arms/groups are evaluated day 2 postoperatively to measure any difference between the two skin closure methods. A high score is used as indicator of traumaticity towards the skin and a higher potential for wound infection.
Time Frame: At postop. day 2 (2 days after kidney donation)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tissue Glue Wound Closure | Conventional Suture + Dressing
Number analyzed (Participants) | 32 | 32
units on a scale | 0 (0) | 0.156 (0.507)

11. Primary Outcome: Wound Healing by Numerical Scales for Blisters Postoperative Day 4.
Description: as for outcome 10
Time Frame: At postop. day 4 (4 days after kidney donation)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tissue Glue Wound Closure | Conventional Suture + Dressing
Number analyzed (Participants) | 32 | 32
units on a scale | 0 (0) | 0.200 (0.542)

12. Primary Outcome: Wound Healing by Numerical Scales for Blisters at Discharge From Hospital.
Description: as for outcome 10
Time Frame: At departure from Surgical Dep. to the patients home, usually at postop. day 4, 5, 6 or 7
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tissue Glue Wound Closure | Conventional Suture + Dressing
Number analyzed (Participants) | 32 | 32
units on a scale | 0 (0) | 0.028 (0.115)

13. Primary Outcome: Wound Healing by Numerical Scales for Gaps Postoperative Day 2.
Description: The evaluation is performed by the use of a previously set numerical scale for gaps (0: no gap - 3: need for resuture/strips). Both arms/groups are evaluated day 2 postoperatively to measure any difference between the two skin closure methods. A high score is used as indicator of traumaticity towards the skin and a higher potential for wound infection.
Time Frame: Postop. day 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tissue Glue Wound Closure | Conventional Suture + Dressing
Number analyzed (Participants) | 32 | 32
units on a scale | 0.094 (0.522) | 0 (0)

14. Primary Outcome: Wound Healing by Numerical Scales for Gaps Postoperative Day 4.
Description: as for outcome 13
Time Frame: Postop. day 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tissue Glue Wound Closure | Conventional Suture + Dressing
Number analyzed (Participants) | 32 | 32
units on a scale | 0.344 (0.888) | 0 (0)

15. Primary Outcome: Wound Healing by Numerical Scales for Gaps at Discharge From Hospital.
Description: as for outcome 13
Time Frame: At departure from Surgical Dep. to the patients home, usually at postop. day 4, 5, 6 or 7
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tissue Glue Wound Closure | Conventional Suture + Dressing
Number analyzed (Participants) | 32 | 32
units on a scale | 0.400 (0.917) | 0 (0)

16. Primary Outcome: TIme Consumption
Description: The specific time required for skin closure (tissue adhesive versus suture) was recorded, counted from initial application of adhesive/intracutaneous suture until final dressing.
Time Frame: The specific time required for skin closure (tissue adhesive versus suture) was recorded, counted from initial application of adhesive/intracutaneous suture until final dressing.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Tissue Glue Wound Closure | Conventional Suture + Dressing
Number analyzed (Participants) | 32 | 32
minutes | 5.832 (1.785) | 8.594 (2.253)

17. Primary Outcome: Patients´Self Satisfaction.
Description: The patients' self-satisfaction was evaluated by means of a questionnaire rating the following 3 domains on a numerical (1-5) scale:
  * Total satisfaction regarding wound healing/wound care. 1 (satisfied) to 5 (dissatisfied)
  * Satisfaction regarding wound discomfort; pain, itching, paresthesia, pressure etc. 1 (almost no discomfort) to 5 (lot of discomfort)
  * Satisfaction regarding wound care; suppleness, practicability versus mobilization, showering etc. 1 (almost no practical challenges) to 5 (lot of practical challenges)
  Patients' Self Satisfaction score was the sum of three domains, ranges from 3 (completely satisfied) to 15 (completely dissatisfied).
  These data were collected at the day of discharge, with guidance from two interviewers.
Time Frame: These data were collected at the day of discharge from hospital (postoperative day 4-8).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tissue Glue Wound Closure | Conventional Suture + Dressing
Number analyzed (Participants) | 32 | 32
units on a scale | 4.968 (1.531) | 4.875 (1.996)

ADVERSE EVENTS:
Arm/Group | Conventional Suture + Dressing | Tissue Glue Wound Closure
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/32
Other Adverse Events (participants affected / at risk) | 0/32 | 0/32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No